CLINICAL TRIAL: NCT03542487
Title: Integration of Blood Glucose Monitoring Into Electronic Health Records
Brief Title: Blood Glucose Monitoring in Electronic Health Records
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Inova Health Care Services (Other)
Collaborators: University of California, Berkeley (Other); Abdul Latif Jameel Poverty Action Lab (Other); General Services Administration (GSA) (U.S. Federal Agency); Department of Health and Human Services (U.S. Federal Agency)
Responsible Party: Sponsor
Allocation: Randomized | Model: Factorial | Masking: None | Purpose: Prevention
Other Study IDs: 17-2642; Project Code: 1729 (Other: General Services Administration (OES))
Record Dates: First submitted 2018-05-15; First posted 2018-05-31 (Actual); Results first posted 2024-09-19 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-05

CONDITIONS: Diabetes Mellitus
Keywords: Self Monitoring of Blood Glucose; Electronic Medical Records; Nudge; Secure Messaging; Behavioral Economics
MeSH Terms: conditions — Diabetes Mellitus

STUDY DESIGN:
Intervention Model Description: Primary care practices will be assigned to a provider-side treatment (physician orientation) or to control. Within treatment assigned practices, individual patients will be assigned to one of four reminder messaging groups (one of which is no messaging).
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (5):
- 1: Control (No Intervention): A randomly selected half of primary care practices in the study sample at Inova Health Care Services will not receive any intervention and patients/physicians located at these practices will continue with business as usual.
- 2a: Practice Orientation- No Reminder (Experimental): In the other randomly selected half of primary care practices in the study sample at Inova Health Care Services, practices will be encouraged to batch order blood glucose flowsheets for all patients with diabetes with active MyChart accounts. The research team will contact physicians and practice managers with an explanation of the initiative and instructions for completing batch orders and viewing entries through the system. Additionally, providers will be given a template for a secure smart-text message to send to all patients receiving the flowsheets, instructing them to enter data for the study period. The secure message will also provide them with information on how to enter data, and on the benefits of tracking blood glucose. Of this group of practices, patients will be divided at the individual level into 4 reminder groups. Arm 2a will receive no additional reminder messaging to enter glucose measurements in the electronic flowsheets.
  Interventions: Behavioral: Practice Orientation
- 2b: Practice Orientation- Standard Reminder (Experimental): Practices will be encouraged to batch order blood glucose flowsheets for all patients with diabetes with active MyChart accounts. The research team will contact physicians and practice managers with an explanation of the initiative and instructions for completing batch orders and viewing entries through the system. Additionally, providers will be given a template for a secure smart-text message to send to all patients receiving the flowsheets, instructing them to enter data for the study period. The secure message will also provide them with information on how to enter data, and on the benefits of tracking blood glucose. Of this group of practices, patients will be divided at the individual level into 4 reminder groups. Arm 2b will receive generic biweekly reminders, addressed from Inova Medical Group, to enter glucose measurements in the electronic flowsheets.
  Interventions: Behavioral: Practice Orientation; Behavioral: Standard Reminder
- 2c: Practice Orientation- Gift Card Reminder (Experimental): Practices will be encouraged to batch order blood glucose flowsheets for all patients with diabetes with active MyChart accounts. The research team will contact physicians and practice managers with an explanation of the initiative and instructions for completing batch orders and viewing entries through the system. Additionally, providers will be given a template for a secure smart-text message to send to all patients receiving the flowsheets, instructing them to enter data for the study period. The secure message will also provide them with information on how to enter data, and on the benefits of tracking blood glucose. Of this group of practices, patients will be divided at the individual level into 4 reminder groups. Arm 2c will receive generic biweekly reminders to enter data, addressed from Inova Medical Group, that will also notify that the patient will be entered to win a $50 gift card for each day entering data.
  Interventions: Behavioral: Practice Orientation; Behavioral: Gift Card Reminder
- 2d: Practice Orientation- Physician Reminder (Experimental): Practices will be encouraged to batch order blood glucose flowsheets for all patients with diabetes with active MyChart accounts. The research team will contact physicians and practice managers with an explanation of the initiative and instructions for completing batch orders and viewing entries through the system. Additionally, providers will be given a template for a secure smart-text message to send to all patients receiving the flowsheets, instructing them to enter data for the study period. The secure message will also provide them with information on how to enter data, and on the benefits of tracking blood glucose. Of this group of practices, patients will be divided at the individual level into 4 reminder groups. Arm 2d will receive biweekly reminders, addressed from their physician, encouraging them to enter glucose measurements in the electronic flowsheets (Note that though messages will be addressed from physician, they will be sent by Inova IT).
  Interventions: Behavioral: Practice Orientation; Behavioral: Physician Reminders

INTERVENTIONS:
Behavioral: Practice Orientation — Practices will be encouraged to batch order blood glucose flowsheets for all patients with diabetes with active MyChart accounts. This will allow diabetic patients at these practices to enter any self-monitored glucose measurements. The research team will contact physicians and practice managers with an explanation of the initiative and instructions for completing batch orders and viewing entries through the system. Additionally, providers will be given a template for a secure smart-text message to send to all patients receiving the flowsheets, instructing them to enter data for the study period. The secure message will also provide them with information on how to enter data, and on the benefits of tracking blood glucose.
  Arms: 2a: Practice Orientation- No Reminder; 2b: Practice Orientation- Standard Reminder; 2c: Practice Orientation- Gift Card Reminder; 2d: Practice Orientation- Physician Reminder
Behavioral: Standard Reminder — Patients receive generic biweekly reminders, addressed from Inova Medical Group, to enter glucose measurements in the electronic flowsheets
  Arms: 2b: Practice Orientation- Standard Reminder
Behavioral: Gift Card Reminder — Patients receive generic biweekly reminders, addressed from Inova Medical Group, to enter glucose measurements in the electronic flowsheets. In these reminders, they will also be notified that that they will be entered to win a $50 gift card for each day entering data.
  Arms: 2c: Practice Orientation- Gift Card Reminder
Behavioral: Physician Reminders — Patients receive biweekly reminders, addressed from their physician, encouraging them to enter glucose measurements in the electronic flowsheets (Note that though messages will be addressed from physician, they will be sent by Inova IT)
  Arms: 2d: Practice Orientation- Physician Reminder

SUMMARY:
This multi-site randomized tral aims to test methods of increasing adoption and integration of blood glucose monitoring into electronic medical records, and to measure the impact of wide-scale adoption on health status of patients with diabetes. To investigate determinants of adoption, the research will combine and test doctor and patient focused approaches to encouraging patient use of blood glucose flow sheets through the online patient portal, MyChart. Adoption will be measured on both the extensive and intensive margin: the number of patients who enter data into the flowsheets at all during the study period, and the mean number of entries per patient during the study period. Conditional on statistically significant increases in adoption, the study will examine corresponding intent-to-treat effects on patient A1c, and consider other indicators of possible mechanisms through which A1c improves or does not improve.

ELIGIBILITY:
Inclusion Criteria:

* Adult patients of Inova physicians at primary care sites other than Ashburn II Primary Care, Lake Ridge Primary Care and Springfield Primary Care
* Current diabetes mellitus diagnosis
* Active MyChart account at time of treatment administration

Exclusion Criteria:

* Patients who participating physicians identify as pregnant
* Patients who participating physicians identify as having contraindications for tracking of blood glucose

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 7052 (Actual)
Dates: Start 2018-05-01 (Actual); Primary Completion 2018-10-31 (Actual); Study Completion 2018-10-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Allyson B Root, MS, Principal Investigator — General Services Administration, UC Berkeley; Season Majors, MSN,RN, Principal Investigator — Inova Health Care Services; Mary Ann Friesen, PhD, Principal Investigator — Inova Health Care Services; Christopher P Connolly, MD, Principal Investigator — Inova Health Care Services
Locations (1):
- Inova Heath System, Falls Church, Virginia, United States

IPD SHARING:
Plan to Share IPD: Undecided

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 20 primary care practices were randomly assigned to treatment (10 practices, 3411 patients) and control (10 practices, 3641 patients). Participants at treated primary care practices whose providers placed flow sheet orders (2182 patients total) were assigned to 1 of 4 reminder message groups to encourage utilization of the flow sheets. Assignment to reminder groups was determined alphabetically by the first letter of participant's last name.
Units Other Than Participants: primary care practices
Groups:
- Experimental: Participants at treated primary care practices whose doctors placed flow sheet orders (2182 patients total) were assigned to 1 of 4 reminder message groups to encourage utilization of the flow sheets
- 2a: Participants in the Practice Orientation- No Reminder: Participants assigned to this group will receive no additional reminder messaging to enter glucose measurements in the electronic flowsheets.
- 2b: Participants in the Practice Orientation- Standard Reminder: Participants in this group will receive generic biweekly reminders, addressed from Inova Medical Group, to enter glucose measurements in the electronic flowsheets
- 2c: Participants in the Practice Orientation- Gift Card Reminder: Participants in this group will receive generic biweekly reminders to enter data, addressed from Inova Medical Group, that will also notify that the patient will be entered to win a $50 gift card for each day entering data.
- 2d: Participants in the Practice Orientation- Physician Reminder: Participants in this group will receive biweekly reminders, addressed from their physician, encouraging them to enter glucose measurements in the electronic flowsheets (Note that though messages will be addressed from physician, they will be sent by Inova IT).
Period: Primary Care Practices Randomization
Arm/Group | 1: Control | Experimental | 2a: Participants in the Practice Orientation- No Reminder | 2b: Participants in the Practice Orientation- Standard Reminder | 2c: Participants in the Practice Orientation- Gift Card Reminder | 2d: Participants in the Practice Orientation- Physician Reminder
Started | 3641; 10 primary care practices | 3411; 10 primary care practices | 0; 0 primary care practices | 0; 0 primary care practices | 0; 0 primary care practices | 0; 0 primary care practices
Completed | 3641; 10 primary care practices | 2182; 10 primary care practices (Participants whose providers ordered flowsheets will be assigned to 1 of 4 treatment group during the next period.) | 0; 0 primary care practices | 0; 0 primary care practices | 0; 0 primary care practices | 0; 0 primary care practices
Not Completed | 0; 0 primary care practices | 1229; 0 primary care practices | 0; 0 primary care practices | 0; 0 primary care practices | 0; 0 primary care practices | 0; 0 primary care practices
Period: Participant Randomization
Arm/Group | 1: Control | Experimental | 2a: Participants in the Practice Orientation- No Reminder | 2b: Participants in the Practice Orientation- Standard Reminder | 2c: Participants in the Practice Orientation- Gift Card Reminder | 2d: Participants in the Practice Orientation- Physician Reminder
Started (Participants assigned to the ten (10) primary care practices in the experimental group, whose providers placed flow sheet orders (totaling 2182 participants), were allocated to one of four reminder message groups. Allocation to these reminder groups was determined alphabetically by the first letter of the participants' last names.) | 0; 0 primary care practices | 0; 0 primary care practices | 466; 10 primary care practices | 589; 10 primary care practices | 554; 10 primary care practices | 573; 10 primary care practices
Completed (Primary care practices in the experimental group were excluded as they did not have any participants with the corresponding first letter of the last names used for participant assignment.) | 0; 0 primary care practices | 0; 0 primary care practices | 466; 8 primary care practices | 589; 7 primary care practices | 554; 7 primary care practices | 573; 7 primary care practices
Not Completed | 0; 0 primary care practices | 0; 0 primary care practices | 0; 2 primary care practices | 0; 3 primary care practices | 0; 3 primary care practices | 0; 3 primary care practices

BASELINE CHARACTERISTICS:
Groups:
- 2b: Participants in the Practice Orientation- Standard Reminder; 2c: Participants in the Practice Orientation- Gift Card Reminder: Participants in this group will receive generic biweekly reminders to enter data, addressed from Inova Medical Group, that will also notify that the patient will be entered to win a $50 gift card for each day entering data.
- Total: Total of all reporting groups
Arm/Group | 1: Control | 2a: Participants in the Practice Orientation- No Reminder | 2b: Participants in the Practice Orientation- Standard Reminder | 2c: Participants in the Practice Orientation- Gift Card Reminder | 2d: Participants in the Practice Orientation- Physician Reminder | Total
Number analyzed (Participants) | 3641 | 762 | 895 | 866 | 888 | 7052
Age, Continuous [Mean (Standard Deviation); unit: years] | 58.863 (14.0) | 58.885 (14.9) | 58.434 (14.7) | 58.756 (14.5) | 59.760 (14.7) | 58.910 (14.3)
Sex/Gender, Customized [Count of Participants; unit: Participants]
  Male | 1958 | 412 | 494 | 478 | 496 | 3838
  Female | 1683 | 350 | 401 | 388 | 392 | 3214
Race/Ethnicity, Customized [Count of Participants; unit: Participants] — Race/Ethnicity reported as Hispanic; White, Non-Hispanic; or Other, Unknown or not Reported due to limitations in the data available to report. Data available for analyses is dependent on information available in the Electronic Medical Records (EMR) and the technical limitations of extracting and compiling datasets from the EMR. Missing, unknown, or multiple ethnicity values were not distinguishable due the limitations and are reported as one combined category.
  Participants
    Ethnicity: Hispanic | 253 | 27 | 62 | 50 | 27 | 419
    Ethnicity: White, Non-Hispanic | 2908 | 622 | 688 | 704 | 743 | 5665
    Ethnicity: Other, Unknown, or Not reported | 480 | 113 | 145 | 112 | 118 | 968
Percent A1c, Baseline [Mean (Standard Deviation); unit: Percent A1c] — Percent A1c represents average blood sugar levels as determined by Hemoglobin A1c (HbA1c) test Population: Data reported only for participants with available A1c test results in their Electronic Medical Record (EMR) during appropriate timeframe.
  Participants with no test results or with missing values in their EMR at appropriate timepoint were not included in analysis.
  Percent A1c
    number analyzed (Participants) | 3483 | 715 | 842 | 825 | 850 | 6715
    (all) | 7.219 (1.587) | 7.327 (2.870) | 7.150 (1.543) | 7.189 (1.600) | 7.168 (1.606) | 7.212 (1.784)

OUTCOME MEASURES:

1. Primary Outcome: Count of Participants Entering Flowsheet Data During Measurement Period, Extensive Margin
Description: Count of participants that entered data to an electronic glucose flowsheet during the measurement period (Count of participants determined with a binary aggregation method; 1= Participant used Flow Sheet at least once during measurement period; 0= Participant did not use Flow Sheet during Measurement Period)
Time Frame: (1-14) weeks after initial practice orientation
Measure: Count of Participants; unit: Participants
Groups:
- 2a: Practice Orientation- No Reminder: Participants assigned to this group will receive no additional reminder messaging to enter glucose measurements in the electronic flowsheets.
- 2b: Practice Orientation- Standard Reminder: Participants in this group will receive generic biweekly reminders, addressed from Inova Medical Group, to enter glucose measurements in the electronic flowsheets
- 2c: Practice Orientation- Gift Card Reminder: Participants in this group will receive generic biweekly reminders to enter data, addressed from Inova Medical Group, that will also notify that the patient will be entered to win a $50 gift card for each day entering data.
- 2d: Practice Orientation- Physician Reminder: Participants in this group will receive biweekly reminders, addressed from their physician, encouraging them to enter glucose measurements in the electronic flowsheets (Note that though messages will be addressed from physician, they will be sent by Inova IT).
Arm/Group | 1: Control | 2a: Practice Orientation- No Reminder | 2b: Practice Orientation- Standard Reminder | 2c: Practice Orientation- Gift Card Reminder | 2d: Practice Orientation- Physician Reminder
Number analyzed (Participants) | 3641 | 762 | 895 | 866 | 888
Participants | 4 | 27 | 44 | 43 | 50

2. Primary Outcome: Participant A1c Test Results (as Percent A1c) at 26 Weeks
Description: Percent A1c represents average blood sugar levels as determined by Hemoglobin A1c (HbA1c) test.
  The HbA1c test measures what percentage of hemoglobin proteins in blood are glycated.
  The most recent and available HbA1c test value (percent A1c) in electronic medical records at appropriate time period was used.
Time Frame: 26 weeks after initial practice orientation
Population: Data reported only for participants with available A1c test results in their Electronic Medical Record (EMR) during appropriate timeframe.
  Participants with no test results or with missing values in their EMR at appropriate timepoint were not included in analysis.
Measure: Mean (Standard Deviation); unit: Percent A1c
Arm/Group | 1: Control | 2a: Practice Orientation- No Reminder | 2b: Practice Orientation- Standard Reminder | 2c: Practice Orientation- Gift Card Reminder | 2d: Practice Orientation- Physician Reminder
Number analyzed (Participants) | 3259 | 675 | 784 | 765 | 803
Percent A1c | 7.179 (1.540) | 7.327 (2.894) | 7.110 (1.474) | 7.227 (1.623) | 7.227 (1.731)

3. Secondary Outcome: Count of Participants Entering Flowsheet Data During Measurement Period, Extensive Margin
Description: as for outcome 1
Time Frame: Beginning of week 15 to 26 weeks after initial practice orientation
Measure: Count of Participants; unit: Participants
Arm/Group | 1: Control | 2a: Practice Orientation- No Reminder | 2b: Practice Orientation- Standard Reminder | 2c: Practice Orientation- Gift Card Reminder | 2d: Practice Orientation- Physician Reminder
Number analyzed (Participants) | 3641 | 762 | 895 | 866 | 888
Participants | 4 | 15 | 17 | 20 | 30

4. Secondary Outcome: Number of Days Participant Used Flowsheet, Intensive
Description: The total number of days of participant use of the electronic glucose flowsheet during the measurement period.
  A day of Participant use of electronic glucose flowsheet is defined here as as day (24 hours) in which the participant performed an entry into an electronic glucose flowsheet.
Time Frame: (1-14); (15-26) weeks after initial practice orientation
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 1: Control | 2a: Practice Orientation- No Reminder | 2b: Practice Orientation- Standard Reminder | 2c: Practice Orientation- Gift Card Reminder | 2d: Practice Orientation- Physician Reminder
Number analyzed (Participants) | 3641 | 762 | 895 | 866 | 888
days
  Weeks 1-14 | 0.011 (0.439) | 0.501 (4.281) | 0.350 (2.693) | 0.663 (5.031) | 0.691 (4.683)
  Weeks 15-26 | 0.009 (0.386) | 0.353 (3.986) | 0.213 (2.865) | 0.406 (4.338) | 0.502 (4.830)

5. Secondary Outcome: Count of Participants With an Open Physician Order for Electronic Glucose Flowsheet
Description: Count of participants that have an open physician order for electronic glucose flowsheet end of the measurement period (Count of participants determined with a binary aggregation method; 1= Participant had an open physician order for electronic Glucose Flow Sheet at end of measurement period; 0= Participant did not have an open physician order for electronic Glucose Flow Sheet at end of measurement period)
Time Frame: at 14 and 26 weeks after initial practice orientation
Measure: Count of Participants; unit: Participants
Arm/Group | 1: Control | 2a: Practice Orientation- No Reminder | 2b: Practice Orientation- Standard Reminder | 2c: Practice Orientation- Gift Card Reminder | 2d: Practice Orientation- Physician Reminder
Number analyzed (Participants) | 3641 | 762 | 895 | 866 | 888
Participants
  Week 14 | 5 | 466 | 589 | 554 | 573
  Week 26 | 6 | 466 | 589 | 555 | 573

6. Secondary Outcome: Number of Days Since Last HbA1c Test
Description: The total number of days that elapsed since participant last had and HbA1c test.
  The number of days was measured by the number of days that passed from the date of the most recent HbA1c test in the Electronic Medical Record and the date of the data extraction at the specified time point.
Time Frame: 14; 26 weeks after initial practice orientation
Population: Data reported only for participants with available A1c test results in their Electronic Medical Record (EMR) during appropriate timeframe.
  Participants with no test results in their EMR at appropriate timepoint were not included in analysis
Measure: Mean (Standard Deviation); unit: days
Arm/Group | 1: Control | 2a: Practice Orientation- No Reminder | 2b: Practice Orientation- Standard Reminder | 2c: Practice Orientation- Gift Card Reminder | 2d: Practice Orientation- Physician Reminder
Number analyzed (Participants) | 3352 | 698 | 801 | 794 | 821
days
  Week 14 | 196.369 (201.15) | 196.828 (205.93) | 205.607 (213.98) | 192.341 (192.651) | 210.748 (216.562)
  Week 26: number analyzed (Participants) | 3259 | 676 | 786 | 768 | 803
  Week 26 | 196.434 (207.394) | 208.781 (215.284) | 216.949 (220.655) | 202.957 (206.877) | 216.812 (229.550)

7. Secondary Outcome: Participant A1c Test Results (as Percent A1c) at 14 Weeks
Description: as for outcome 2
Time Frame: 14 weeks after initial practice orientation
Population: as for outcome 2
Measure: Mean (Standard Deviation); unit: Percent A1c
Arm/Group | 1: Control | 2a: Practice Orientation- No Reminder | 2b: Practice Orientation- Standard Reminder | 2c: Practice Orientation- Gift Card Reminder | 2d: Practice Orientation- Physician Reminder
Number analyzed (Participants) | 3351 | 698 | 800 | 792 | 821
Percent A1c | 7.196 (1.601) | 7.276 (2.823) | 7.123 (1.465) | 7.183 (1.593) | 7.197 (1.767)

8. Secondary Outcome: Count of Participants With Improvement of HbA1c Test Results
Description: Count of participants with improved HbA1c test result values in most recent Electronic Medical Record (EMR) during measurement period as compared to HbA1c test value at baseline. (Count of participants determined with a binary aggregation method; 1= Participant Improved, most recent A1c test value less than baseline A1c test value; 0= Participant did not Improve; most recent A1c test value greater than or equal to baseline A1c test value)
  Improvement of HbA1c test results is defined as a reduction of the most recent and available HbA1c test value (a lower percent A1c) in the EMR at appropriate time period relative to the baseline.
  Percent A1c represents average blood sugar levels as determined by Hemoglobin A1c (HbA1c) test The HbA1c test measures what percentage of hemoglobin proteins in blood are glycated.
  Higher percent A1c levels are associated with poor blood sugar control and increased risk of of diabetes-related complications.
Time Frame: 14; 26 weeks after initial practice orientation
Population: Data reported only for participants with available A1c test results in their Electronic Medical Record (EMR) during appropriate timeframes.
  Participants with no test results or with missing values in their EMR at appropriate timepoints were not included in analysis.
Measure: Count of Participants; unit: Participants
Arm/Group | 1: Control | 2a: Practice Orientation- No Reminder | 2b: Practice Orientation- Standard Reminder | 2c: Practice Orientation- Gift Card Reminder | 2d: Practice Orientation- Physician Reminder
Number analyzed (Participants) | 3333 | 693 | 796 | 790 | 818
Participants
  At Week 14 | 666 | 155 | 158 | 160 | 147
  At Week 26: number analyzed (Participants) | 3232 | 669 | 778 | 759 | 798
  At Week 26 | 961 | 195 | 229 | 204 | 215

9. Secondary Outcome: Count of Participants With Percent A1c Below Benchmark of 7
Description: Count of participants with most recent HbA1c test value (percent A1c) in Electronic Medical Records below target benchmark of 7 at appropriate time point (Count of participants determined with a binary aggregation method; 1= Participant HbA1c test value less than 7; 0= Participant Hb1Ac test value greater than or equal to 7).
  Percent A1c represents average blood sugar levels as determined by Hemoglobin A1c (HbA1c) test.
  The HbA1c test measures what percentage of hemoglobin proteins in blood are glycated.
  A percent A1c level less than 7 is a common treatment target and is associated with with a lower risk of diabetes-related complications.
Time Frame: 14; 26 weeks after initial practice orientation
Population: as for outcome 2
Measure: Count of Participants; unit: Participants
Arm/Group | 1: Control | 2a: Practice Orientation- No Reminder | 2b: Practice Orientation- Standard Reminder | 2c: Practice Orientation- Gift Card Reminder | 2d: Practice Orientation- Physician Reminder
Number analyzed (Participants) | 3351 | 698 | 800 | 792 | 821
Participants
  At Week 14 | 1846 | 388 | 453 | 442 | 458
  At Week 26: number analyzed (Participants) | 3259 | 675 | 784 | 765 | 803
  At Week 26 | 1799 | 368 | 453 | 421 | 443

10. Secondary Outcome: Total Secure Messages Sent by Participant
Description: Total number of messages sent by participant via MyChart Electronic medical records system during the measurement period
Time Frame: (1-14); (15-26) weeks after initial practice orientation
Measure: Mean (Standard Deviation); unit: number of messages
Arm/Group | 1: Control | 2a: Practice Orientation- No Reminder | 2b: Practice Orientation- Standard Reminder | 2c: Practice Orientation- Gift Card Reminder | 2d: Practice Orientation- Physician Reminder
Number analyzed (Participants) | 3641 | 762 | 895 | 866 | 888
number of messages
  Weeks 1-14 | 1.385 (3.016) | 1.407 (2.872) | 1.528 (3.272) | 1.434 (2.638) | 1.571 (3.282)
  Weeks 15-26 | 1.128 (2.65) | 1.226 (2.803) | 1.077 (2.496) | 1.037 (2.338) | 1.135 (2.597)

11. Secondary Outcome: Total Secure Messages Sent by Patient to Primary Care Provider
Description: Total number of MyChart messages sent by patient to the Primary Care Provider (PCP) during the measurement period. Not reported separately from Total number of messages sent by patient, so outcomes not reported here.
Time Frame: (1-14); (15-26) weeks after initial practice orientation
Population: Data not collected.
Arm/Group | 1: Control | 2a: Practice Orientation- No Reminder | 2b: Practice Orientation- Standard Reminder | 2c: Practice Orientation- Gift Card Reminder | 2d: Practice Orientation- Physician Reminder
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

12. Secondary Outcome: Total Secure Messages Sent by PCP to Patient
Description: Total number of MyChart messages sent by PCP to the patient during the measurement period
Time Frame: (1-14); (15-26) weeks after initial practice orientation
Population: Data not collected.
Arm/Group | 1: Control | 2a: Practice Orientation- No Reminder | 2b: Practice Orientation- Standard Reminder | 2c: Practice Orientation- Gift Card Reminder | 2d: Practice Orientation- Physician Reminder
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

13. Secondary Outcome: Total Number of Participant Phone Appointments
Description: Total number of participant phone appointments during the measurement period
Time Frame: (1-14); (1-26) weeks after initial practice orientation
Measure: Mean (Standard Deviation); unit: number of phone appointments
Arm/Group | 1: Control | 2a: Practice Orientation- No Reminder | 2b: Practice Orientation- Standard Reminder | 2c: Practice Orientation- Gift Card Reminder | 2d: Practice Orientation- Physician Reminder
Number analyzed (Participants) | 3641 | 762 | 895 | 866 | 888
number of phone appointments
  Weeks 1-14 | 0.792 (1.651) | 0.827 (1.64) | 0.789 (1.613) | 0.849 (1.654) | 0.765 (1.432)
  Weeks 1-26 | 1.442 (2.547) | 1.457 (2.417) | 1.398 (2.506) | 1.485 (2.525) | 1.434 (2.420)

14. Secondary Outcome: Total Number of Participant In-person Appointments
Description: Total number of participant in-person appointments during the measurement period
Time Frame: (1-14); (1-26) weeks after initial practice orientation
Measure: Mean (Standard Deviation); unit: number of appointments
Arm/Group | 1: Control | 2a: Practice Orientation- No Reminder | 2b: Practice Orientation- Standard Reminder | 2c: Practice Orientation- Gift Card Reminder | 2d: Practice Orientation- Physician Reminder
Number analyzed (Participants) | 3641 | 762 | 895 | 866 | 888
number of appointments
  Weeks 1-14 | 1.275 (3.476) | 1.314 (3.914) | 1.251 (3.580) | 1.109 (2.782) | 1.191 (2.991)
  Weeks 1-26 | 2.326 (5.322) | 2.358 (5.4) | 2.153 (4.775) | 2.083 (4.652) | 2.188 (4.452)

15. Secondary Outcome: Count of Participants With Changes to Active Medication List
Description: Count of Participants with Changes (Any; Addition; Removal) to list of active medications in EMR during measurement period. Active medication lists is comprised of prescription ordered medications for participants.
  Count of participants determined with a binary aggregation method:
  Any Change is defined as medications added or removed from active list ( 1= Participant had medications added to or removed from active medication list; 0= Participant did not have medication added to or removed from active medication list).
  Medications Added is defined as the addition of medications to active medication list ( 1= Participant had medications added to active medication list; 0= Participant did not have medications added to active medication list).
  Medications Removed is defined as the removal of medications to active medication list ( 1= Participant had medications removed from active medication list; 0= Participant did not have medications removed from active medication list).
Time Frame: (1-14); (1-26) weeks after initial practice orientation
Measure: Count of Participants; unit: Participants
Arm/Group | 1: Control | 2a: Practice Orientation- No Reminder | 2b: Practice Orientation- Standard Reminder | 2c: Practice Orientation- Gift Card Reminder | 2d: Practice Orientation- Physician Reminder
Number analyzed (Participants) | 3641 | 762 | 895 | 866 | 888
Participants
  Any Change - Weeks 1-14 | 742 | 135 | 133 | 141 | 140
  Any Change - Weeks 1-26 | 1132 | 198 | 199 | 223 | 251
  Medication Added - Weeks 1-14 | 709 | 129 | 131 | 137 | 137
  Medication Added - Weeks 1-26 | 1087 | 188 | 188 | 214 | 247
  Medication Removed - Weeks 1-14 | 395 | 71 | 73 | 75 | 77
  Medication Removed - Weeks 1-26 | 555 | 96 | 95 | 117 | 121

16. Secondary Outcome: Prescription Orders
Description: Number of prescription ordered medications for participant during measurement period (Total all; Total new/non-refill; Total diabetes related)
Time Frame: (1-14); (1-26) weeks after initial practice orientation
Measure: Mean (Standard Deviation); unit: number of orders
Arm/Group | 1: Control | 2a: Practice Orientation- No Reminder | 2b: Practice Orientation- Standard Reminder | 2c: Practice Orientation- Gift Card Reminder | 2d: Practice Orientation- Physician Reminder
Number analyzed (Participants) | 3641 | 762 | 895 | 866 | 888
number of orders
  Number of Total Prescription Orders - Weeks 1-14 | 5.111 (19.825) | 5.912 (19.041) | 4.488 (13.612) | 4.733 (18.286) | 4.259 (12.866)
  Number of Total Prescription Orders - Weeks 1-26 | 9.296 (32.904) | 10.554 (33.799) | 8.050 (22.783) | 8.242 (31.365) | 7.795 (20.211)
  Number of Non-Refill Orders - Weeks 1-14 | 5.111 (19.825) | 5.192 (19.041) | 4.488 (13.612) | 4.733 (18.286) | 4.259 (12.866)
  Number of Non-Refill Orders - Weeks 1-26 | 9.296 (32.904) | 10.544 (33.799) | 8.050 (22.783) | 8.242 (31.365) | 7.795 (20.211)
  Number of Diabetes Related Prescription Orders - Weeks 1-14 | 0.678 (2.218) | 0.718 (1.686) | 0.591 (1.605) | 0.691 (1.749) | 0.574 (1.335)
  Number of Diabetes Related Prescription Orders - Weeks 1-26 | 1.28 (3.592) | 1.318 (2.938) | 1.036 (2.311) | 1.162 (2.756) | 1.063 (2.055)

17. Secondary Outcome: Flowsheet Entry Values (Descriptive)
Description: Value of blood glucose entered into flowsheet (descriptive analysis). No systematic outcomes recorded to report.
Time Frame: 2; 4; 6; 8; 10; 12; 14; 18; 22; 26 weeks after initial orientation meeting
Population: Data not collected.
Arm/Group | 1: Control | 2a: Practice Orientation- No Reminder | 2b: Practice Orientation- Standard Reminder | 2c: Practice Orientation- Gift Card Reminder | 2d: Practice Orientation- Physician Reminder
Number analyzed (Participants) | 0 | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Description: Death, serious adverse events, and other (non-serious adverse events) were not assessed for this study.
Arm/Group | 1: Control | 2a: Practice Orientation- No Reminder | 2b: Practice Orientation- Standard Reminder | 2c: Practice Orientation- Gift Card Reminder | 2d: Practice Orientation- Physician Reminder
All-Cause Mortality (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Serious Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0
Other Adverse Events (participants affected / at risk) | 0/0 | 0/0 | 0/0 | 0/0 | 0/0

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2019-02-21): https://cdn.clinicaltrials.gov/large-docs/87/NCT03542487/Prot_SAP_001.pdf